CLINICAL TRIAL: NCT03411902
Title: Effect of Bisphosphonate Use on Surgical Weight Loss Associated Bone Loss in Older Adults With Morbid Obesity
Brief Title: Weight Loss With Risedronate for Bone Health
Acronym: WERISE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Wake Forest University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00048310
Record Dates: First submitted 2018-01-11; First posted 2018-01-26 (Actual); Results first posted 2021-01-22 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2020-12

CONDITIONS: Bariatric Surgery Candidate; Bone Loss; Weight Loss
Keywords: Bone Health
MeSH Terms: conditions — Bone Diseases, Metabolic; Weight Loss | interventions — Risedronic Acid

STUDY DESIGN:
Intervention Model Description: This pilot study is a RCT, involving 24 sleeve gastrectomy patients randomized to Risedronate or placebo capsules for 24 weeks
Who Masked: Participant, Care Provider
Masking Description: Both participant and research associate charged with administering medication or placebo capsules will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Risedronate (Active Comparator): Experimental: Risedronate sodium,150 mg capsule once every 4 weeks for 24 weeks.
  Interventions: Drug: Risedronate Sodium 150 MG
- Placebo (Placebo Comparator): Active comparator: Identical 150 mg placebo capsules once every 4 weeks for 24 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Risedronate Sodium 150 MG — Subjects randomized to the Risedronate group will take a 150 mg capsule of oral Risedronate once every 4 weeks for 24 weeks (6 doses), beginning 1 week prior to surgery and dispensed in blinded capsules from the WFSM research pharmacy.
  Other Names: Code A
  Arms: Risedronate
Other: Placebo — Participants randomized to the placebo group will receive 150 mg placebo capsule once every 4 weeks for 24 weeks (6 doses), beginning 1 week prior to surgery and dispensed in blinded capsules from the WFSM research pharmacy.
  Other Names: Code B
  Arms: Placebo

SUMMARY:
This is a pilot project to determine the feasibility of recruiting, enrolling, treating, and following 24 older sleeve gastrectomy patients into a randomized controlled trial (RCT) examining the efficacy of bisphosphonate use versus placebo in the prevention of surgical weight loss associated loss of bone mass and quality.

DETAILED DESCRIPTION:
This pilot study is a RCT, involving 24 participants randomized to Risedronate or placebo capsules for 24 weeks. All subjects planning a sleeve gastrectomy (SG) procedure will be approached during their pre-surgical evaluation for possible participation in the study. Eligible participants will be referred onto the study coordinator to read/sign an IRB-approved informed consent prior to enrollment.

Two in-person baseline assessment visits [baseline visit 1 (BV1), baseline visit 2 (BV2)] occurring 1-6 weeks prior to surgery, and two in-person follow up assessment visits [follow up visit 1 (FV1) and follow up visit 2 (FV2)] occurring ±2 weeks from their 23-week post-surgery date will be conducted, as well as monthly medication compliance reminders and adverse event reporting via phone. Optional additional exploratory assessments include CT-derive bone health and blood-based biomarkers, as well as 12-month DXA, CT, and blood assessments. The Wake Forest WMC, under the direction of Drs. Ard and Fernandez, will serve as a source of recruitment for potential study participants.

ELIGIBILITY:
Inclusion Criteria

* Subjects planning a sleeve gastrectomy procedure
* 40-79 yrs of age
* Willingness to provide informed consent
* Agreement to all study procedures and assessments

Exclusion Criteria

* Age <40 years
* Baseline weight >450 pounds
* Chronic anti-reflux treatment
* History of medical disorders known to affect bone metabolism
* Use of bone-active medications
* Known allergy to Risedronate

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male and female
Enrollment: 24 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen M Beavers, PhD, Principal Investigator — Wake Forest University
Locations (1):
- Wake Forest University, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Swafford AA, Ard JD, Beavers DP, Gearren PC, Fernandez AZ, Ford SA, Greene KA, Kammire DE, Nesbit BA, Reed KK, Weaver AA, Beavers KM. Risedronate to Prevent Bone Loss After Sleeve Gastrectomy: Study Design and Feasibility Report of a Pilot Randomized Controlled Trial. JBMR Plus. 2020 Oct 2;4(10):e10407. doi: 10.1002/jbm4.10407. eCollection 2020 Oct. PMID 33103032

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Risedronate | Placebo
Started | 11 | 13
Completed | 8 | 13
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Risedronate | Placebo | Total
Number analyzed (Participants) | 11 | 13 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (7.7) | 57.3 (5.7) | 55.7 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 3 | 2 | 5
  White | 8 | 11 | 19
Region of Enrollment [Number; unit: participants]
  United States | 11 | 13 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Enrolled Participants That Completed All 24 Week Procedures
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Risedronate | Placebo
Number analyzed (Participants) | 11 | 13
Participants | 8 | 13

2. Secondary Outcome: Fat Pounds
Description: Duel-energy x-ray absorptiometry (DXA)-Acquired Measure--Fat pounds portion of Total body composition
Time Frame: 24 weeks
Population: 3 subjects were lost to follow up in the risedronate arm
Measure: Mean (95% Confidence Interval); unit: pounds
Arm/Group | Risedronate | Placebo
Number analyzed (Participants) | 8 | 13
pounds | 45.6 [41.8 to 49.4] | 40.6 [37.9 to 43.4]
Statistical Analysis 1: Comparison: Risedronate vs Placebo; Test type: Superiority; p = 0.048, Mixed Models Analysis

3. Secondary Outcome: Lean Pounds
Description: Duel-energy x-ray absorptiometry (DXA)-Acquired Measure--Lean pounds portion of Total body composition
Time Frame: 24 weeks
Population: 3 subjects were lost to follow up in the risedronate arm
Measure: Mean (95% Confidence Interval); unit: pounds
Arm/Group | Risedronate | Placebo
Number analyzed (Participants) | 8 | 13
pounds | 50.4 [49.1 to 51.8] | 50.7 [49.7 to 51.7]
Statistical Analysis 1: Comparison: Risedronate vs Placebo; Test type: Superiority; p = 0.745, Mixed Models Analysis

4. Secondary Outcome: Total Change in Femoral Neck Hip Density
Description: Duel-energy x-ray absorptiometry (DXA)-Acquired Measure for Total Hip Density measured in g/cm^2
Time Frame: Baseline and 24 weeks
Population: Three subjects were lost to follow up in the risedronate arm.
Measure: Mean (95% Confidence Interval); unit: g/cm^2
Arm/Group | Risedronate | Placebo
Number analyzed (Participants) | 8 | 13
g/cm^2 | -0.028 [-0.049 to -0.006] | -0.047 [-0.063 to -0.030]
Statistical Analysis 1: Comparison: Risedronate vs Placebo; Test type: Superiority; p = 0.163, Mixed Models Analysis

5. Secondary Outcome: Total Change in Lumbar Spine Density
Description: Duel-energy x-ray absorptiometry (DXA)-Acquired Measure for Lumbar Spine Density measured in g/cm^2
Time Frame: Baseline and 24 weeks
Population: Three subjects were lost to follow up in the risedronate arm.
Measure: Mean (95% Confidence Interval); unit: g/cm^2
Arm/Group | Risedronate | Placebo
Number analyzed (Participants) | 8 | 13
g/cm^2 | 0.028 [-0.006 to 0.063] | -0.029 [-0.054 to -0.004]
Statistical Analysis 1: Comparison: Risedronate vs Placebo; Test type: Superiority; p = 0.013, Mixed Models Analysis

6. Secondary Outcome: Duel-energy X-ray Absorptiometry (DXA)-Acquired Measure for Ultradistal Radius (or UD Radius) Density
Description: Total change in ultradistal radius density measure in g/cm^2
Time Frame: 24 weeks
Population: Three subjects were lost to follow up in the risedronate arm.
Measure: Mean (95% Confidence Interval); unit: g/cm^2
Arm/Group | Risedronate | Placebo
Number analyzed (Participants) | 8 | 13
g/cm^2
  Radius 33 BMD (g/cm^2) | -0.002 [-0.027 to 0.023] | -0.016 [-0.036 to 0.004]
  Radius UD BMD (g/cm^2) | 0.000 [-0.017 to 0.017] | -0.013 [-0.026 to 0.001]
Statistical Analysis 1: Comparison: Risedronate vs Placebo; Pertaining to Radius 33 BMD; Test type: Superiority; p = 0.337, Mixed Models Analysis
Statistical Analysis 2: Comparison: Risedronate vs Placebo; Pertaining to Radius UD BMD; Test type: Superiority; p = 0.238, Mixed Models Analysis

7. Secondary Outcome: Trabecular Bone Score (TBS)
Description: TBS of the lumbar spine measured by two dimensional (2D) variogram acquired through duel-energy x-ray absorptiometry (DXA). Trabecular bone score is a unitless index of bone microarchitecture. A high TBS value means that bone microarchitecture is dense and well connected, with little space between trabeculae. The following normal range for TBS values in postmenopausal women has been proposed: TBS >=1.350 is considered to be normal; TBS between 1.200 and 1.350 is considered to be consistent with partially degraded microarchitecture; and TBS <=1.200 defines degraded microarchitecture
Time Frame: 24 weeks
Population: Three subjects were lost to follow up in the risedronate arm.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Risedronate | Placebo
Number analyzed (Participants) | 8 | 13
score on a scale | 1.478 [1.413 to 1.543] | 1.485 [1.436 to 1.533]
Statistical Analysis 1: Comparison: Risedronate vs Placebo; Test type: Superiority; p = 0.860, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: baseline through 12 months
Arm/Group | Risedronate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/13
Other Adverse Events (participants affected / at risk) | 4/11 | 3/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risedronate (N=11) | Placebo (N=13)
thyroid cancer (Endocrine disorders) | 1 (1) | 0 (0)
melanoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risedronate (N=11) | Placebo (N=13)
headache (Nervous system disorders) | 0 (0) | 1 (1)
psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
gastroesophageal reflux disease exacerbation (Gastrointestinal disorders) | 0 (0) | 1 (1)
broken ankle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Broken humerus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Informed Consent Form (2020-06-02): https://cdn.clinicaltrials.gov/large-docs/02/NCT03411902/ICF_000.pdf
  • Study Protocol (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT03411902/Prot_001.pdf
  • Statistical Analysis Plan (2020-12-29): https://cdn.clinicaltrials.gov/large-docs/02/NCT03411902/SAP_002.pdf